CLINICAL TRIAL: NCT02066402
Title: A Phase 3 Randomized, Double-Blind, Multicenter Study Comparing the Efficacy and Safety of Intravenous to Oral 6-Day Tedizolid Phosphate and Intravenous to Oral 10-Day Linezolid for the Treatment of Acute Bacterial Skin and Skin Structure Infections
Brief Title: Efficacy and Safety of Intravenous to Oral 6-Day Tedizolid Phosphate vs. Intravenous to Oral 10-Day Linezolid in Patients With Acute Bacterial Skin and Skin Structure Infection (ABSSSI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16121
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — tedizolid; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tedizolid Phosphate (Sivextro, BAY119-2631) (Experimental): Participants received 200 mg Tedizolid Phosphate once daily intravenous (I.V.) infusion to oral for 6 days, followed by 4 days of placebo.
  Interventions: Drug: Tedizolid (BAY119-2631); Drug: Placebo Tedizolid (BAY119-2631); Drug: Placebo Linezolid
- Linezolid (Active Comparator): Participants received 600 mg Linezolid twice daily I.V. infusion to oral for 10 days.
  Interventions: Drug: Placebo Tedizolid (BAY119-2631); Drug: Linezolid

INTERVENTIONS:
Drug: Tedizolid (BAY119-2631) — 50 % of the participants will be randomized to this arm and will receive 200 mg Tedizolid once daily i.v to oral from 1-6 days
  Arms: Tedizolid Phosphate (Sivextro, BAY119-2631)
Drug: Placebo Tedizolid (BAY119-2631) — 50 % of the participants will be randomized to this arm and will receive 200 mg Placebo Tedizolid once daily i.v to oral from 7-10 days
Drug: Linezolid — 50 % of the participants will be randomized to this arm and will receive 600 mg Linezolid twice daily i.v. to oral from 1-10 days
  Arms: Linezolid
Drug: Placebo Linezolid — 50 % of the participants will be randomized to this arm and will receive 600 mg Placebo Linezolid twice daily i.v. to oral from 1-10 days
  Arms: Tedizolid Phosphate (Sivextro, BAY119-2631)

SUMMARY:
This study is aimed to evaluate the efficacy and safety between Tedizolid 200mg daily (intra venous) I.V. to oral for 6-day treatment compared with that of Linezolid 600mg twice daily I.V. to oral for 10-day treatment Acute Bacterial Skin and skin structure infection (ABSSSI).This is a double-blind, randomized, active control, 7-10days treatment for all subjects.

DETAILED DESCRIPTION:
Number of participants with adverse evnets as a measure of safety and tolerability will be covered in Adverse Events section.

ABSSSI Efficacy Safety Tedizolid Phosphate Linezolid

ELIGIBILITY:
Inclusion Criteria:

* Males or females >/=18 years old
* Adequate venous access for a minimum of 2 I.V. doses of study drug
* Acute Bacterial Skin and skin structure infection (ABSSSI) meeting at least 1 of the clinical syndrome definitions listed below and requiring I.V. antibiotic therapy. Local symptoms must have started within 7 days before the Screening Visit

  * Cellulitis/erysipelas
  * Major cutaneous abscess
  * Wound Infection
* Suspected or documented gram-positive infection from baseline Gram stain or culture.

Exclusion Criteria:

* Uncomplicated skin and skin structure infections such as furuncles, minor abscesses
* Infections associated with, or in close proximity to, a prosthetic device
* Severe sepsis or septic shock
* Known bacteremia at time of screening
* ABSSSI due to or associated with any of the following:

  * Suspected or documented gram-negative pathogens in patients with cellulitis/erysipelas or major cutaneous abscess that require an antibiotic with specific gram-negative coverage. Patients with wound infections where gram-negative adjunctive therapy is warranted may be enrolled if they meet the other eligibility criteria
  * Diabetic foot infections, gangrene, or perianal abscess
  * Concomitant infection at another site not including a secondary ABSSSI lesion (eg, septic arthritis, endocarditis, osteomyelitis)
  * Infected burns
  * Decubitus or chronic skin ulcer, or ischemic ulcer due to peripheral vascular disease (arterial or venous)
  * Any evolving necrotizing process (ie, necrotizing fasciitis)
* Use of antibiotics as follows:

  * Systemic antibiotic with gram-positive cocci activity for the treatment of any infection within 24 hours before the first infusion of study drug
  * Patients who failed prior therapy for the primary infection site are also excluded from enrollment
  * Topical antibiotic on the primary lesion within 24 hours before the first infusion of study drug except for antibiotic/antiseptic-coated dressing applied to the clean postsurgical wound
* Administration of Linezolid within 30 days before the first infusion of the study drug
* Recent history of opportunistic infections where the underlying cause of these infections is still active (eg, leukemia, transplant, acquired immunodeficiency syndrome [AIDS])
* Previous exposure to Tedizolid Phosphate treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2014-03-04 (Actual); Primary Completion 2016-03-06 (Actual); Study Completion 2016-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (34):
- United States (5):
  - Chula Vista, California
  - La Mesa, California
  - Oceanside, California
  - Las Vegas, Nevada
  - Teaneck, New Jersey
- China (22):
  - Wuhu, Anhui
  - Fuzhou, Fujian
  - Guangzhou, Guangdong
  - Wuhan, Hubei
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Suzhou, Jiangsu
  - Wuxi, Jiangsu
  - Changchun, Jilin
  - Dalian, Liaoning
  - Shenyang, Liaoning
  - Xi'an, Shaanxi
  - Jinan, Shandong
  - Taiyuan, Shanxi
  - Chengdu, Sichuan
  - Ürümqi, Xinjiang
  - Kunming, Yunnan
  - Hangzhou, Zhejiang
  - Beijing
  - Chongqing
  - Shanghai
  - Tianjin
- Philippines (2):
  - City of Taguig
  - Quezon City
- Taiwan (5):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District

REFERENCES:
- [Derived] Lv X, Alder J, Li L, O'Riordan W, Rybak MJ, Ye H, Zhang R, Zhang Z, Zhu X, Wilcox MH. Efficacy and Safety of Tedizolid Phosphate versus Linezolid in a Randomized Phase 3 Trial in Patients with Acute Bacterial Skin and Skin Structure Infection. Antimicrob Agents Chemother. 2019 Jun 24;63(7):e02252-18. doi: 10.1128/AAC.02252-18. Print 2019 Jul. PMID 30988146

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid
Started | 300 | 298
Participants Received Treatment | 292 | 297
Completed Study Treatment Period | 261 | 256
Completed | 274 | 275
Not Completed | 26 | 23
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 11 | 8
Not completed — Withdrawal by Subject | 14 | 11
Not completed — Progressive disease-clinical progression | 0 | 1
Not completed — Protocol driven decision point | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid | Total
Number analyzed (Participants) | 300 | 298 | 598
Age, Customized [Number; unit: Participants]
  < 65 years | 259 | 245 | 504
  65 - 75 years | 33 | 35 | 68
  > 75 years | 8 | 18 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 106 | 197
  Male | 209 | 192 | 401
Visual analog scale (VAS) pain scores [Mean (Standard Deviation); unit: Units on a scale] — The patient-reported level of pain were assessed by the visual analog scale (VAS) pain score. VAS pain score ranged from 0 mm (no pain) to 100 mm (worst pain ever). It used a 100 mm VAS to instruct the patient to indicate the point along the line that represents the pain they are feeling. Once the patient indicates how much pain they are feeling, measure the distance from no pain and enter the value.
  Units on a scale | 53.2 (27.3) | 53.9 (28.7) | 53.6 (28.0)
Wong-Baker faces rating scale (FRS) pain scores [Mean (Standard Deviation); unit: Units on a scale] — The patient-reported level of pain were assessed by the faces rating scale (FRS) pain score. Ask the patient to rate their pain from 0 to 10 with 0 being no pain at all and 10 being the worst pain then enter the numerical value.
  Units on a scale | 5.6 (2.6) | 5.7 (2.7) | 5.6 (2.7)
Type of acute bacterial skin and skin structure infections (ABSSSI) infection [Number; unit: Participants]
  Cellulitis/erysipelas | 192 | 191 | 383
  Major cutaneous abscess | 40 | 39 | 79
  Wound infection | 68 | 68 | 136

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Early Clinical Response at 48-72 Hours After the First Infusion of Study Drug in the ITT Analysis Set.
Description: Early clinical response is defined as responder if there is >=20% reduction in the area of erythema, edema, and/or induration (length × width) of the primary acute bacterial skin and skin structure infections (ABSSSI) lesion, compared with baseline at the 48-72 Hour visit.
Time Frame: Baseline and 48-72 hours visit
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid
Number analyzed (Participants) | 300 | 298
Percentage of participants | 75.3 | 79.9
Statistical Analysis 1: Comparison: Tedizolid Phosphate (Sivextro, BAY119-2631) vs Linezolid; Test type: Non-Inferiority or Equivalence — The non-inferiority (NI) hypothesis test is a 1-sided hypothesis test performed at the 2.5% level of significance. Predefined margin for non-inferiority is -10%; p = 0.2027, Fisher Exact; Difference of responder rate = -4.6, 95% CI 2-sided [-11.2 to 2.2]

2. Secondary Outcome: Programmatically Defined Clinical Response at End of Therapy (EOT) Visit in the ITT Analysis Set
Description: Clinical Failure: Presence of fever; No lesion size decrease from baseline; Clinician assessment of tenderness worse than mild; Persistent same or great intensity purulent drainage of wound infection; Confounding use of systemic concomitant antibiotic; TEAE lead to study drug discontinuation; Require additional antibiotic treatment for primary lesion; Unplanned major surgical intervention. Clinical Success: Afebrile or fever due to other cause; Lesion size decrease from baseline; Clinician assessment of mild/absent tenderness; None/lesser intensity purulent drainage of wound infection; None confounding use of systemic concomitant antibiotic; None TEAE leading to study drug discontinuation; No additional antibiotic therapy for primary lesion; No unplanned major surgical intervention; No osteomyelitis after baseline; For wound/abscess: no incision/drainage of the ABSSSI site after Day1 unless planned. For cellulitis/ersipelas: no incision/drainage of the ABSSSI site after 48-72 H Visit.
Time Frame: Baseline and EOT visit (Day 11)
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid
Number analyzed (Participants) | 300 | 298
Percentage of participants
  Clinical success | 82.0 | 84.2
  Clinical failure or Indeterminate | 18.0 | 15.8
Statistical Analysis 1: Comparison: Tedizolid Phosphate (Sivextro, BAY119-2631) vs Linezolid; Test type: Non-Inferiority or Equivalence — The non-inferiority (NI) hypothesis test is a 1-sided hypothesis test performed at the 2.5% level of significance; Difference of responder rate = -2.2, 95% CI 2-sided [-8.3 to 3.8]

3. Secondary Outcome: Programmatically Defined Clinical Response at End of Therapy (EOT) Visit in the Clinically Evaluable at EOT (CE-EOT) Analysis Set
Description: Clinical response will be defined as percentage of participants with clinical success, clinical failure or indeterminate.
Time Frame: Baseline and EOT visit (Day 11)
Population: CE-EOT
Measure: Number; unit: Percentage of participants
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid
Number analyzed (Participants) | 242 | 243
Percentage of participants
  Clinical success | 89.7 | 91.8
  Clinical failure or Indeterminate | 10.3 | 8.2
Statistical Analysis 1: Comparison: Tedizolid Phosphate (Sivextro, BAY119-2631) vs Linezolid; Test type: Non-Inferiority or Equivalence — The non-inferiority (NI) hypothesis test is a 1-sided hypothesis test performed at the 2.5% level of significance; Difference of responder rate = -2.1, 95% CI 2-sided [-7.4 to 3.2]

4. Secondary Outcome: Overall Investigator's Assessment of Clinical Success at Post Therapy Evaluation (PTE) Visit (7-14 Days After EOT Visit) in the ITT Analysis Set
Description: The Investigator made an assessment of clinical response at the PTE Visit (7-14 days after the EOT Visit +2 days). Participants assessed as a clinical failure at the EOT Visit are considered a clinical failure at the PTE Visit. Percentage of participants with clinical success, clinical failure or indeterminate were reported.
Time Frame: Baseline and post-therapy evaluation visit (7-14 days after Day 11)
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid
Number analyzed (Participants) | 300 | 298
Percentage of participants
  Clinical success | 79.7 | 81.9
  Clinical failure or Indeterminate | 20.3 | 18.1
Statistical Analysis 1: Comparison: Tedizolid Phosphate (Sivextro, BAY119-2631) vs Linezolid; Test type: Non-Inferiority or Equivalence — The non-inferiority (NI) hypothesis test is a 1-sided hypothesis test performed at the 2.5% level of significance; Difference of responder rate = -2.2, 95% CI 2-sided [-8.6 to 4.1]

5. Secondary Outcome: Overall Investigator's Assessment of Clinical Success at Post Therapy Evaluation (PTE) Visit (7-14 Days After EOT Visit) in the Clinically Evaluable at Post Therapy Evaluation (CE-PTE) Analysis Set
Description: as for outcome 4
Time Frame: Baseline and post-therapy evaluation visit (7-14 days after Day 11)
Population: CE-PTE
Measure: Number; unit: Percentage of participants
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid
Number analyzed (Participants) | 219 | 231
Percentage of participants
  Clinical success | 90.4 | 93.5
  Clinical failure or Indeterminate | 9.6 | 6.5
Statistical Analysis 1: Comparison: Tedizolid Phosphate (Sivextro, BAY119-2631) vs Linezolid; Test type: Non-Inferiority or Equivalence — The non-inferiority (NI) hypothesis test is a 1-sided hypothesis test performed at the 2.5% level of significance; Difference of responder rate = -3.1, 95% CI 2-sided [-8.4 to 2.0]

6. Secondary Outcome: Investigator's Assessment of Clinical Response at 48-72 Hours
Description: The Investigator made an assessment of clinical response at the 48-72 Hour Visit based on following definition: Improving (Improvement in overall clinical status of ABSSSI compatible with continuation of study drug therapy); Stable (Signs and symptoms stable, no apparent change in overall clinical status but compatible with continuation of study drug therapy); Other.
Time Frame: Baseline and at 48-72 hours
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid
Number analyzed (Participants) | 300 | 298
Percentage of participants
  Improving | 86.7 | 90.3
  Stable | 4.7 | 3.0
  Other | 0.7 | 0.0
  Missing | 8.0 | 6.7

7. Secondary Outcome: Investigator's Assessment of Clinical Response at Day 7 Visit
Description: The Investigator made an assessment of clinical response at Day 7 Visit based on following definition: Improving (Improvement in overall clinical status of ABSSSI compatible with continuation of study drug therapy); Other.
Time Frame: Baseline and Day 7 visit
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid
Number analyzed (Participants) | 300 | 298
Percentage of participants
  Improving | 88.3 | 87.6
  Other | 0.3 | 0.3
  Missing | 11.3 | 12.1

8. Secondary Outcome: Value of the Visual Analog Scale (VAS) Pain Scores at Each Time Point
Description: The patient-reported level of pain were assessed by the visual analog scale (VAS) pain score. VAS pain score ranged from 0 mm (no pain) to 100 mm (worst pain ever). It used a 100 mm VAS to instruct the patient to indicate the point along the line that represents the pain they are feeling. Once the patient indicates how much pain they are feeling, measure the distance from no pain and enter the value.
Time Frame: Up to EOT visit (Day 11)
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid
Number analyzed (Participants) | 300 | 298
Units on a scale
  Day 2 | 40.9 (26.3) | 40.1 (26.5)
  48-72 hours | 30.2 (25.6) | 30.7 (25.7)
  Day 7 | 18.8 (22.9) | 17.8 (21.2)
  EOT | 11.6 (19.4) | 10.3 (18.1)

9. Secondary Outcome: Change From Baseline in the Visual Analog Scale (VAS) Pain Scores at Each Time Point
Description: as for outcome 8
Time Frame: Up to EOT visit (Day 11)
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid
Number analyzed (Participants) | 300 | 298
Units on a scale
  Day 2 | -12.5 (21.7) | -13.8 (20.1)
  48-72 hours | -23.2 (23.9) | -23.2 (24.3)
  Day 7 | -34.7 (26.7) | -36.1 (26.7)
  EOT | -41.6 (28.3) | -43.6 (29.1)

10. Secondary Outcome: Value of the Faces Rating Scale (FRS) Pain Scores at Each Time Point
Description: The patient-reported level of pain were assessed by the faces rating scale (FRS) pain score. Ask the patient to rate their pain from 0 to 10 with 0 being no pain at all and 10 being the worst pain then enter the numerical value.
Time Frame: Up to EOT visit (Day 11)
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid
Number analyzed (Participants) | 300 | 298
Units on a scale
  Day 2 | 4.1 (2.4) | 4.2 (2.5)
  48-72 hours | 3.2 (2.4) | 3.2 (2.5)
  Day 7 | 2.1 (2.3) | 2.0 (2.2)
  EOT | 1.3 (2.0) | 1.3 (1.9)

11. Secondary Outcome: Change From Baseline in the Faces Rating Scale (FRS) Pain Scores at Each Time Point
Description: The patient-reported level of pain were assessed by the faces rating scale (FRS) pain score. The patient-reported level of pain were assessed by the faces rating scale (FRS) pain score. Ask the patient to rate their pain from 0 to 10 with 0 being no pain at all and 10 being the worst pain then enter the numerical value.
Time Frame: Up to EOT visit (Day 11)
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid
Number analyzed (Participants) | 300 | 298
Units on a scale
  Day 2 | -1.5 (2.0) | -1.5 (1.8)
  48-72 hours | -2.4 (2.2) | -2.4 (2.3)
  Day 7 | -3.5 (2.6) | -3.6 (2.5)
  EOT | -4.2 (2.8) | -4.4 (2.7)

ADVERSE EVENTS:
Time Frame: From the start of study drug administration until last subject last visit.
Arm/Group | Tedizolid Phosphate (Sivextro, BAY119-2631) | Linezolid
Serious Adverse Events (participants affected / at risk) | 11/292 | 8/297
Other Adverse Events (participants affected / at risk) | 60/292 | 63/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tedizolid Phosphate (Sivextro, BAY119-2631) (N=292) | Linezolid (N=297)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0
Therapeutic product ineffective (General disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 4
Erysipelas (Infections and infestations) | 2 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Infected bite (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tedizolid Phosphate (Sivextro, BAY119-2631) (N=292) | Linezolid (N=297)
Diarrhoea (Gastrointestinal disorders) | 7 | 8
Nausea (Gastrointestinal disorders) | 15 | 14
Fatigue (General disorders) | 3 | 6
Injection site extravasation (General disorders) | 5 | 6
Pyrexia (General disorders) | 10 | 5
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 7
Cellulitis (Infections and infestations) | 7 | 9
Skin bacterial infection (Infections and infestations) | 6 | 7
Alanine aminotransferase increased (Investigations) | 7 | 6
Aspartate aminotransferase increased (Investigations) | 7 | 6
Dizziness (Nervous system disorders) | 3 | 7
Headache (Nervous system disorders) | 6 | 7
Phlebitis (Vascular disorders) | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less